CLINICAL TRIAL: NCT05153226
Title: Graft vs Host Disease Prophylaxis in Unrelated Donor Transplantation: a Randomized Clinical Trial Comparing PTCY vs ATG (GRAPPA)
Brief Title: GvHD Prophylaxis in Unrelated Donor HCT: Randomized Trial Comparing PTCY Versus ATG
Acronym: GRAPPA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: DKMS gemeinnützige GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DKMS-21-01; 2021-000853-17 (EudraCT Number)
Record Dates: First submitted 2021-11-26; First posted 2021-12-10 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Graft Vs Host Disease; Peripheral Blood Stem Cell Transplantation; AML; MDS; MDS/MPN; CMML
Keywords: Graft vs Host Disease; Peripheral Blood Stem Cell Transplantation; Cyclophsophamide; Anti-thymocyte globulin (rabbit)
MeSH Terms: conditions — Graft vs Host Disease | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cyclophosphamide (Experimental): Cyclophosphamide 50 mg/kg (AIBW) i.v. d+3, d+4 post transplant
  Interventions: Drug: Cyclophosphamide
- ATG (Active Comparator): ATG Grafalon 10 mg/kg i.v. d-3, d-2, d-1 pre-transplant
  Interventions: Biological: ATG

INTERVENTIONS:
Drug: Cyclophosphamide — 50 mg/kg (AIBW) i.v. d+3, d+4 post transplant
  Other Names: all brands
  Arms: Cyclophosphamide
Biological: ATG — 10 mg/kg i.v. d-3, d-2, d-1 pre-transplant
  Other Names: ATG Grafalon
  Arms: ATG

SUMMARY:
Post-transplantation cyclophosphamide (PTCY) has become increasingly popular in the haploidentical HCT setting because it overcomes the HLA-mismatch barrier and levels GVHD risk. This advantage may also prove useful in the context of unrelated donor (UD) transplantation. GVHD prophylaxis for matched unrelated donor hematopoietic cell transplantation (alloHCT) in Europe is mainly conducted with ATG. Still, the burden of acute and chronic GVHD and especially of relapse remains high with both approaches for GVHD prevention.

PTCY has not been tested against the current standard ATG for GvHD prophylaxis in large randomized trials. The goal of this trial is to compare the outcomes of PTCY and ATG for patients receiving unrelated donor PBSCT. PTCY-based prophylaxis promises to have beneficial net effects on immune reconstitution, GVHD and disease control, and thus might impact on patient survival.

ELIGIBILITY:
Inclusion Criteria:

* Signed written Informed Consent and able to understand the nature of the trial and the trial related procedures and to comply with them.
* Age ≥ 18 years.
* One of the following eligible diagnoses: AML in CR1 with intermediate or adverse risk genetic abnormalities (according to the ELN 2017 guidelines), or undefined risk. AML of any ELN risk category after hematological or molecular relapse, or with primary refractory disease. AML arising from myelodysplastic syndrome (MDS) or a myeloproliferative neoplasia, except if favourable genetic abnormalities (according to ELN 2017 guidelines) are present. Therapy-related myeloid neoplasia (t-MN), except if favourable genetic abnormalities (according to ELN 2017 guidelines) are present. MDS with intermediate risk, high risk or very high risk disease (according to the IPSS-R Score) regardless of treatment status. MDS/MPN and CMML-1/CMML-2 regardless of treatment status.
* The left ventricular ejection fraction (LVEF) was assessed ≥40% at last echocardiography.
* Transplantation with Peripheral Blood Stem Cells (PBSC) scheduled to be performed 4 to 14 days after date of randomization.
* The scheduled donor is unrelated to the patient, and matched or partially matched (with not more than one allele or antigen mismatch) at HLA-A, -B, -C, or -DRB1.
* Absence of pregnancy confirmed by highly sensitive pregnancy test for WOCBP. Test must not date back more than 3 days prior to randomization, or more than 3 days prior to start of conditioning, if it started before randomization.

Exclusion Criteria:

* Anamnestic intravenous or subcutaneous exposure to rabbit immunoglobin-preparations (e.g. Grafalon or Thymoglobulin)
* Known hypersensitivity to ATG-Grafalon or its excipients.
* Known hypersensitivity to cyclophosphamide, its metabolites or excipients.
* Prior allogeneic hematopoietic transplantation.
* Patients who receive supplementary continuous oxygen at the time of randomization.
* Symptomatic heart failure (NYHA ≥2) at the time of randomization.
* Uncontrolled viral, bacterial or fungal infection with progression or no clinical improvement at the time of randomization.
* Symptomatic cystitis or known obstruction of urine flow at the time of randomization.
* Breast-feeding women.
* WOCBP and fertile male patients unable or unwilling to follow highly effective contraception methods from enrollment to minimum six months after the last dose of the IMP.
* Simultaneous participation in another interventional clinical trial with an investigational medicinal product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | from randomization
GVHD- and relapse-free survival (GRFS) | from HCT

SECONDARY OUTCOMES:
Overall survival | from HCT
Relapse- and immunosuppression-free survival (RIFS) | from HCT
Event-free survival | 1 year
Cumulative incidence of relapse | 1 year
Cumulative incidence of non-relapse mortality | 1 year
Cumulative incidences of acute and chronic GVHD | 180 days and 2 years after HCT

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Schetelig, Prof Dr med, Study Chair — Universitätsklinikum Dresden
Locations (23):
- Germany (23):
  - Uniklinik RWTH Aachen, Aachen
  - Univeristätsklinikum Augsburg, Augsburg
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Universitätsklinikum Köln, Cologne
  - St.-Johannes-Hospital Dortmund, Dortmund
  - Universitätsklinikum Dresden, Dresden
  - Uniklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Essen (AöR), Essen
  - Universitätsklinikum Frankfurt, Frankfurt am Main
  - Universitätsklinikum Halle (Saale), Halle
  - Universitätsklinikum des Saarlandes, Homburg
  - Universitätsklinikum Jena, Jena
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Universitätsmedizin Mainz, Mainz
  - Universitätsmedizin Mannheim, Mannheim
  - Philipps Universität Marburg, Marburg
  - Universitätsklinikum Münster, Münster
  - Klinikum Nürnberg Nord, Nuremberg
  - Universitätsmedizin Rostock, Rostock
  - Robert-Bosch-Krankenhaus, Stuttgart
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinikum Würzburg, Würzburg